CLINICAL TRIAL: NCT03043313
Title: MOUNTAINEER: A Phase II, Open Label Study of Tucatinib Combined With Trastuzumab in Patients With HER2+ Metastatic Colorectal Cancer
Brief Title: Tucatinib Plus Trastuzumab in Patients With HER2+ Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Academic and Community Cancer Research United (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGNTUC-017; NCI-2017-01107 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACCRU-GI-1617 (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2017-01-31; First posted 2017-02-06 (Estimated); Results first posted 2023-04-18 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Colorectal Adenocarcinoma
Keywords: HER2; ERBB2; Colorectal cancer; Seattle Genetics
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trastuzumab; tucatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Tucatinib + Trastuzumab (Experimental): Non-randomized cohort. Participants take tucatinib twice per day orally on Days 1-21 and trastuzumab intravenously (into the vein; IV) on Day 1. Cycles repeat every 21 days.
  Interventions: Drug: Trastuzumab; Drug: Tucatinib
- Cohort B: Tucatinib + Trastuzumab (Experimental): Randomized cohort. Participants take tucatinib twice per day orally on Days 1-21 and trastuzumab intravenously (into the vein; IV) on Day 1. Cycles repeat every 21 days.
  Interventions: Drug: Trastuzumab; Drug: Tucatinib
- Cohort C: Tucatinib Monotherapy (Experimental): Randomized cohort. Participants take tucatinib twice per orally every day. Participants who do not respond to therapy may have the option to receive tucatinib and trastuzumab.
  Interventions: Drug: Tucatinib

INTERVENTIONS:
Drug: Trastuzumab — Given intravenously (into the vein; IV)
  Other Names: Herceptin
  Arms: Cohort A: Tucatinib + Trastuzumab; Cohort B: Tucatinib + Trastuzumab
Drug: Tucatinib — Given orally
  Other Names: ARRY-380; ONT-380; TUKYSA

SUMMARY:
This trial studies how well the drug tucatinib works when given with trastuzumab and when given by itself. The participants in this trial have HER2-positive (HER2+) metastatic colorectal cancer (mCRC). 'Metastatic' means that the cancer has spread to other parts of the body.

In the first part of this study, participants enrolled into Cohort A and received both tucatinib and trastuzumab. In the second part of this study, participants are randomly assigned to either Cohort B or Cohort C. Participants in Cohort B will receive tucatinib and trastuzumab. Participants in Cohort C will receive tucatinib. Participants in Cohort C who do not respond to therapy may have an option to receive tucatinib plus trastuzumab.

ELIGIBILITY:
Inclusion Criteria

* Histologically and/or cytologically documented adenocarcinoma of the colon or rectum that is metastatic and/or unresectable
* Unless contraindicated, participants must have received and failed regimens containing the following agents: fluoropyrimidine (e.g., 5-fluorouracil or capecitabine), oxaliplatin, irinotecan, an anti-VEGF monoclonal antibody (bevacizumab, ramucirumab, or ziv-aflibercept), and an anti-PD-(L)1 therapy (nivolumab or pembrolizumab) if tumor has deficient mismatch repair proteins or is MSI-High.
* Have progression of unresectable or metastatic CRC after the last systemic therapy, or be intolerant of last systemic therapy
* Have RAS wild-type in primary or metastatic tumor tissue, based on expanded RAS testing
* Willing and able to provide the most recently available tissue blocks obtained prior to treatment initiation. If archival tissue is not available, then a newly-obtained baseline biopsy of an accessible tumor
* Have confirmed HER2-positive mCRC, as defined by having tumor tissue tested at a Clinical Laboratory Improvement Act (CLIA)-certified or International Organization for Standardization (ISO)-accredited laboratory, meeting at least one of the following criteria:

  * HER2+ overexpression (3+ immunohistochemistry [IHC]) by an FDA-approved or Conformité Européene (CE)-marked HER2 ICH test
  * HER2 2+ IHC is eligible if the tumor is amplified by an FDA-approved or CE-marked HER2 in situ hybridization assay (FISH or chromogenic in situ hybridization [CISH]))
  * HER2 (ERBB2) amplification by CLIA-certified or ISO-accredited next generation sequencing (NGS) sequencing assay
* Have radiographically measurable disease assessable by RECIST 1.1, with at least one site of disease that is measurable and that has not been previously irradiated; or, if the participant has had previous radiation to the target lesion(s), there must be evidence of progression since the radiation
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
* Life expectancy greater than 3 months
* Have adequate hematological, hepatic, renal, coagulation, and cardiac function

Exclusion Criteria

* Previous treatment with anti-HER2 targeting therapy
* Previous treatment with any systemic anticancer therapy, non-central nervous system radiation, or experimental agent within 3 weeks of first dose of study treatment
* Toxicity related to prior cancer therapies that has not resolved to ≤ Grade 1, with the following exceptions:

  * Alopecia and neuropathy, which must have resolved to ≤ Grade 2
  * Congestive heart failure (CHF), which must have been ≤ Grade 1 in severity at the time of occurrence, and must have resolved completely
  * Anemia, which must have resolved to ≤ Grade 2
  * Decreased ANC, which must have resolved to ≤ Grade 2
* Have clinically significant cardiopulmonary disease
* Have known myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or cardiac surgery within 6 months prior to first dose of study treatment
* Major surgical procedure, open biopsy, or significant traumatic injury ≤28 days prior to enrollment (≤56 days for hepatectomy, open thoracotomy, or major neurosurgery) or anticipation of need for major surgical procedure during the study
* Serious, non-healing wound, ulcer, or bone fracture
* Known to be positive for hepatitis B by surface antigen expression
* Known to have active hepatitis C infection

  * Exception for participants with a documented sustained virologic response of 12 weeks
* Known to be positive for human immunodeficiency virus (HIV)
* Subjects who are pregnant, breastfeeding, or planning a pregnancy
* Inability to swallow pills or any significant gastrointestinal disease which would preclude the adequate oral absorption of medications
* Have used strong CYP2C8 inhibitor within 5 half-lives of the inhibitor, or have used a strong CYP2C8 or CYP3A4 inducer within 5 days prior to first dose of study treatment
* History of another malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy.

  * Exceptions are malignancies with a negligible risk of metastasis or death
* Subjects with known active CNS metastasis

  * Irradiated or resected lesions are permitted, provided the lesions are fully treated and inactive, subject is asymptomatic, and no steroids have been administered for at least 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2023-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Strickler, Study Chair — Academic and Community Cancer Research United; Jorge Ramos, DO, Study Director — Seagen Inc.
Locations (56):
- United States (41):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Pacific Shores Medical Group, Long Beach, California
  - Keck Medical Center / University of Southern California, Los Angeles, California
  - Cedars Sinai Medical Center / Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - Saint Joseph Heritage Medical Group, Santa Rosa, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Lombardi Cancer Center / Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists - South Region, Fort Myers, Florida
  - Florida Cancer Specialists - North Region, St. Petersburg, Florida
  - Winship Cancer Institute / Emory University School of Medicine, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute / Wayne State University, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University / University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Tennessee Oncology-Nashville/Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology - Beaumont, Beaumont, Texas
  - Texas Oncology - Baylor Sammons Cancer Center, Dallas, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Providence Regional Medical Center Everett, Everett, Washington
  - Seattle Cancer Care Alliance / University of Washington, Seattle, Washington
  - Aurora Research Institute Cancer Center, Milwaukee, Wisconsin
- Belgium (3):
  - Cliniques Universitaires Saint Luc, Brussels, Other
  - Universitair Ziekenhuis Antwerpen, Edegem, Other
  - UZ Leuven campus Gasthuisberg, Leuven, Other
- France (5):
  - Hospitalier Jean Minjoz, Besançon, Other
  - Center Georges Francois Leclerc, Dijon, Other
  - Hôpital Franco-Britannique - Fondation Cognacq-Jay, Levallois-Perret, Other
  - Centre Leon Berard - Centre regional de lutte contre le cancer Rhone-Alpes, Lyon, Other
  - Hopital Saint-Antoine, Paris, Other
- Italy (3):
  - Instituto Europeo di Oncologia, Milan, Other
  - Niguarda Ca' Granda Hospital, Milan, Other
  - Azienda Ospedaliero-Universitaria Pisana - Ospedale S. Chiara, Pisa, Other
- Spain (4):
  - Hospital Universitario Vall d'Hebron, Barcelona, Other
  - Institut Catala d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), L'Hospitalet de Llobregat, Other
  - Hospital General Universitario Gregorio Maranon, Madrid, Other
  - Hospital Clinico Universitario de Valencia, Valencia, Other

REFERENCES:
- [Derived] Zhang D, Taylor A, Zhao JJ, Endres CJ, Topletz-Erickson A. Population Pharmacokinetic Analysis of Tucatinib in Healthy Participants and Patients with Breast Cancer or Colorectal Cancer. Clin Pharmacokinet. 2024 Oct;63(10):1477-1487. doi: 10.1007/s40262-024-01412-0. Epub 2024 Oct 5. PMID 39368039
- [Derived] Strickler JH, Bekaii-Saab TS. A study to learn how well tucatinib plus trastuzumab works for treating participants with metastatic colorectal cancer, and how safe it is: a plain language summary of the MOUNTAINEER study. Future Oncol. 2024 Mar;20(8):409-421. doi: 10.2217/fon-2023-0676. Epub 2023 Nov 8. PMID 37941353
- [Derived] Casak SJ, Horiba MN, Yuan M, Cheng J, Lemery SJ, Shen YL, Fu W, Moore JN, Li Y, Bi Y, Auth D, Fesenko N, Kluetz PG, Pazdur R, Fashoyin-Aje LA. FDA Approval Summary: Tucatinib with Trastuzumab for Advanced Unresectable or Metastatic, Chemotherapy Refractory, HER2-Positive RAS Wild-Type Colorectal Cancer. Clin Cancer Res. 2023 Nov 1;29(21):4326-4330. doi: 10.1158/1078-0432.CCR-23-1041. PMID 37318379
- [Derived] Strickler JH, Cercek A, Siena S, Andre T, Ng K, Van Cutsem E, Wu C, Paulson AS, Hubbard JM, Coveler AL, Fountzilas C, Kardosh A, Kasi PM, Lenz HJ, Ciombor KK, Elez E, Bajor DL, Cremolini C, Sanchez F, Stecher M, Feng W, Bekaii-Saab TS; MOUNTAINEER investigators. Tucatinib plus trastuzumab for chemotherapy-refractory, HER2-positive, RAS wild-type unresectable or metastatic colorectal cancer (MOUNTAINEER): a multicentre, open-label, phase 2 study. Lancet Oncol. 2023 May;24(5):496-508. doi: 10.1016/S1470-2045(23)00150-X. PMID 37142372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 117 participants were enrolled at a total of 56 sites in the United States, Italy, France, Belgium, and Spain. The date of first participant enrollment was 23-Jun-2017. The date of last participant randomization was 02-Nov-2023.
Groups:
- Tucatinib+Trastuzumab (Cohort A): Non-randomized cohort. Participants received Tucatinib 300 milligrams (mg) orally (PO) twice daily (BID) on Days 1 to 21 of each 21-day cycle. Trastuzumab 8 milligram/kilogram (mg/kg) by intravenous (IV) infusion on Day 1 of Cycle 1 and 6 mg/kg on Day 1 of each subsequent cycle until progressive disease (PD), death, withdrawal of consent, study closure, or alternative therapy.
- Tucatinib+Trastuzumab (Cohort B): Randomized cohort. Participants received Tucatinib 300 mg PO BID on Days 1 to 21 of each 21-day cycle. Trastuzumab 8 mg/kg by IV infusion on Day 1 of Cycle 1 and 6 mg/kg on Day 1 of each subsequent cycle until PD, death, withdrawal of consent, study closure, or alternative therapy.
- Tucatinib Monotherapy (Cohort C): Participants received Tucatinib 300 mg PO BID on Days 1 to 21 of each 21-day cycle. Participants who did not respond to monotherapy were given the option to receive tucatinib and trastuzumab until PD, death, withdrawal of consent, study closure, or alternative therapy based on radiographic progression (as determined by investigator assessment using response evaluation criteria in solid tumors [RECIST] version [v] 1.1), or if they had not achieved a partial response (PR) or complete response (CR) by the week 12 assessment.
Period: Overall Study
Arm/Group | Tucatinib+Trastuzumab (Cohort A) | Tucatinib+Trastuzumab (Cohort B) | Tucatinib Monotherapy (Cohort C)
Started | 45 | 41 | 31
Completed | 0 | 0 | 0
Not Completed | 45 | 41 | 31
Not completed — Withdrawal by Subject | 5 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Death | 28 | 26 | 17
Not completed — Participation terminated by sponsor | 11 | 13 | 13

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set included all participants who were enrolled and received any amount of study treatment and had human epidermal growth factor receptor 2+ (HER2+) tumors as defined by one or more protocol required local tests.
Groups:
- Tucatinib+Trastuzumab (Cohort A): Non-randomized cohort. Participants received Tucatinib 300 mg PO BID on Days 1 to 21 of each 21-day cycle. Trastuzumab 8 mg/kg by IV infusion on Day 1 of Cycle 1 and 6 mg/kg on Day 1 of each subsequent cycle until PD, death, withdrawal of consent, study closure, or alternative therapy.
- Tucatinib Monotherapy (Cohort C): Participants received Tucatinib 300 mg PO BID on Days 1 to 21 of each 21-day cycle. Participants who did not respond to monotherapy were given the option to receive tucatinib and trastuzumab until PD, death, withdrawal of consent, study closure, or alternative therapy based on radiographic progression (as determined by investigator assessment using RECIST v1.1), or if they had not achieved a PR or CR by the week 12 assessment.
- Total: Total of all reporting groups
Arm/Group | Tucatinib+Trastuzumab (Cohort A) | Tucatinib+Trastuzumab (Cohort B) | Tucatinib Monotherapy (Cohort C) | Total
Number analyzed (Participants) | 45 | 39 | 30 | 114
Age, Continuous [Median (Full Range); unit: Years] | 52 [24 to 71] | 57 [31 to 77] | 59.5 [29 to 75] | 56 [24 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 15 | 48
  Male | 26 | 25 | 15 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 35 | 29 | 25 | 89
  Unknown or Not Reported | 8 | 9 | 4 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 3 | 6
  White | 37 | 28 | 23 | 88
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 3 | 8 | 4 | 15
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG performance status was used to assess participants disease progression, and ability to carry out daily living activities. 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed less than (<)50 percent (%) of the time; 3= In bed >50% of the time; 4=100% bedridden; 5=Dead.
  Participants
    Grade 0 | 24 | 26 | 17 | 67
    Grade 1 | 20 | 11 | 13 | 44
    Grade 2 | 1 | 2 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 45 | 24 | 16 | 85
  Europe | 0 | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (cORR) Per RECIST v1.1 Per Blinded Independent Central Review (BICR) in Pooled Cohorts A+B
Description: cORR was defined as the percentage of participants with confirmed CR or PR according to RECIST v1.1. CR was defined as the disappearance of all target lesions and each target lymph node must have reduction in short axis to less than (<)1.0 centimeter (cm). PR was defined as at least a 30 percentage (%) decrease in post-baseline sum of the diameters (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the baseline sum of diameters.
Time Frame: Up to 46.6 months
Population: The Full Analysis Set included all participants who were enrolled and received any amount of study treatment and had HER2+ tumors as defined by one or more protocol required local tests. Data for cohort A and B was combined as prespecified in the statistical analysis plan (SAP).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Tucatinib+Trastuzumab (Cohorts A+B): Participants received Tucatinib 300 mg PO BID on Days 1 to 21 of each 21-day cycle. Trastuzumab 8 mg/kg by IV infusion on Day 1 of Cycle 1 and 6 mg/kg on Day 1 of each subsequent cycle until PD, death, withdrawal of consent, study closure, or alternative therapy.
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B)
Number analyzed (Participants) | 84
Percentage of Participants | 39.3 [28.8 to 50.5]

2. Secondary Outcome: ORR by 12 Weeks of Treatment Per RECIST v1.1 According to BICR Assessment
Description: ORR per BICR by 12 Weeks was defined as the percentage of participants with CR or PR by 12 weeks of treatment, and before time of crossover (Cohort C), whichever came earlier. CR was defined as the disappearance of all target lesions and each target lymph node must have reduction in short axis to more than <1.0 cm. PR was defined as at least a 30% decrease in post-baseline sum of the diameters (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the baseline sum of diameter.
Time Frame: Up to 3 months
Population: The Full Analysis Set included all participants who were enrolled and received any amount of study treatment and had HER2+ tumors as defined by one or more protocol required local tests. Data for cohort A and B was combined as prespecified in SAP.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Tucatinib Pre-Crossover (Cohort C): Participants received Tucatinib 300 mg PO BID on Days 1 to 21 of each 21-day cycle. Participants who did not respond to monotherapy were given the option to receive tucatinib and trastuzumab based on radiographic progression (as determined by investigator assessment using RECIST v1.1), or if they had not achieved a PR or CR by the week 12 assessment.
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B) | Tucatinib Pre-Crossover (Cohort C)
Number analyzed (Participants) | 84 | 30
Percentage of Participants | 28.6 [19.2 to 39.5] | 3.3 [0.1 to 17.2]

3. Secondary Outcome: Duration of Response (DOR) Per RECIST v1.1 According to BICR Assessment
Description: DOR was defined as the time from the first objective response (CR or PR that is subsequently confirmed) to documented PD per RECIST v1.1 or death from any cause, whichever occurred first. CR was defined as the disappearance of all target lesions and each target lymph node must have reduction in short axis to more than <1.0 cm. PR was defined as at least a 30% decrease in post-baseline sum of the diameters (PBSD) (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the BSD. PD was defined as: at least one new malignant lesion, which also includes any lymph node that was normal at baseline (<1.0 cm short axis) and increased to more than or equal to (>=)1.0 cm short axis during follow-up or at least a 20% increase in PBSD taking as reference the minimum sum of the diameters (MSD). In addition, the PBSD must also demonstrate an absolute increase of at least 0.5 cm from the MSD.
Time Frame: Up to 64.1 months
Population: The Full Analysis Set included all participants who were enrolled and received any amount of study treatment and had HER2+ tumors as defined by one or more protocol required local tests. Data for cohort A and B was combined as prespecified in SAP. Here, "Number of Participants Analyzed" signifies participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B) | Tucatinib Pre-Crossover (Cohort C)
Number analyzed (Participants) | 33 | 30
Months | 15.2 [8.9 to 20.5] | NA [NA to NA] — Data for median and lower or upper limits could not be estimated due to insufficient participants with event.

4. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST v1.1 According to BICR Assessment for Pooled Cohorts A+B
Description: PFS was defined as the time from start of study treatment (Cohort A) or date of randomization (Cohort B) to documented disease progression (as determined by BICR per RECIST v1.1) or death from any cause, whichever occurred first. PD was defined as: at least one new malignant lesion, which also included any lymph node that was normal at baseline (<1.0 cm short axis) and increased to >=1.0 cm short axis during follow-up or at least a 20% increase in post-baseline sum of the diameters (PBSD) taking as reference the minimum sum of the diameters (MSD). In addition, the PBSD must also demonstrate an absolute increase of at least 0.5 cm from the MSD.
Time Frame: Up to 64.1 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B)
Number analyzed (Participants) | 84
Months | 8.1 [4.2 to 10.2]

5. Secondary Outcome: Overall Survival (OS) in Pooled Cohorts A+B
Description: OS was defined as the time from start of study treatment (Cohort A) or randomization (Cohort B) to date of death due to any cause.
Time Frame: Up to 71.8 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B)
Number analyzed (Participants) | 84
Months | 23.9 [18.7 to 28.3]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs): Interim Analysis
Description: AE: Any untoward medical occurrence in a participant or clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. Treatment emergent AEs (TEAEs): Events that were new or worsened on or after receiving the first dose of study treatment (tucatinib or trastuzumab) and up through 30 days after the last dose of study treatment (tucatinib or trastuzumab). Serious AE (SAE): An event that at any dose led to death; life-threatening; required inpatient hospitalization/prolongation of existing hospitalization; persistent/significant disability/incapacity; congenital anomaly/birth defect/ important medical event. Treatment related AEs, SAEs, deaths also included. Relatedness was judged by investigator According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03: Grade(G) 3=severe AE, G4=life-threatening, urgent intervention indicated, G5=death related to AE.
Time Frame: Up to 49.3 months
Population: The safety analysis set included participants who received any amount of study treatment. Data for cohort A and B was combined as prespecified in SAP.
Measure: Count of Participants; unit: Participants
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B) | Tucatinib Pre-Crossover (Cohort C)
Number analyzed (Participants) | 86 | 30
Participants
  Any TEAE | 82 | 28
  Tucatinib-related TEAE | 63 | 22
  Trastuzumab-related TEAE | 58 | NA — Tucatinib monotherapy arm.
  Any grade 3-5 TEAE | 33 | 8
  Trastuzumab-related grade 3-5 TEAE | 6 | NA — Tucatinib monotherapy arm.
  Tucatinib-related grade 3-5 TEAE | 8 | 2
  Any Treatment-Emergent Serious AE (TESAE) | 19 | 3
  Tucatinib-related TESAE | 3 | 1
  Trastuzumab-related TESAE | 2 | NA — Tucatinib monotherapy arm.
  TEAE leading to death | 0 | 0
  Discontinuation of any study treatment due to TEAE | 5 | 0
  Discontinuation of tucatinib due to TEAE | 5 | 0
  Discontinuation of tucatinib due to tucatinib-related TEAE | 2 | 0
  Discontinuation of trastuzumab due to TEAE | 3 | NA — Tucatinib monotherapy arm.
  Discontinuation of trastuzumab due to trastuzumab-related TEAE | 0 | NA — Tucatinib monotherapy arm.

7. Secondary Outcome: Number of Participants With AEs: Final Analysis
Description: AE: Any untoward medical occurrence in a participant or clinical investigational participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. Treatment emergent AEs (TEAEs): Events that were new or worsened on or after receiving the first dose of study treatment (tucatinib or trastuzumab) and up through 30 days after the last dose of study treatment (tucatinib or trastuzumab). SAE: An event that at any dose led to death; life-threatening; required inpatient hospitalization/prolongation of existing hospitalization; persistent/significant disability/incapacity; congenital anomaly/birth defect/ important medical event. Treatment related AEs, SAEs, deaths also included. Relatedness was judged by investigator According to NCI CTCAE version 4.03: Grade(G) 3=severe AE, G4=life-threatening, urgent intervention indicated, G5=death related to AE.
Time Frame: Up to 65.1 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Groups:
- Tucatinib Post-Crossover (Cohort C): Participants received Tucatinib 300 mg PO BID on Days 1 to 21 of each 21-day cycle. Trastuzumab 8 mg/kg by IV infusion on Day 1 of Cycle 1 and 6 mg/kg on Day 1 of each subsequent cycle until PD, death, withdrawal of consent, study closure, or alternative therapy.
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B) | Tucatinib Post-Crossover (Cohort C)
Number analyzed (Participants) | 86 | 28
Participants
  Any TEAE | 82 | 23
  Tucatinib-related TEAE | 64 | 15
  Trastuzumab-related TEAE | 59 | 13
  More than or equal to (>=) Grade 3 TEAE | 35 | 9
  Tucatinib-related >= grade 3 TEAE | 8 | 2
  Trastuzumab-related >= grade 3 TEAE | 6 | 2
  Any Treatment-Emergent Serious AE (TESAE) | 20 | 6
  Tucatinib-related TESAE | 3 | 0
  Trastuzumab-related TESAE | 2 | 2
  TEAE leading to death | 0 | 0
  Discontinuation of any study treatment due to TEAE | 5 | 2
  Discontinuation of tucatinib due to treatment-related TEAE | 2 | 2
  Discontinuation of tucatinib due to tucatinib-related TEAE | 2 | 2
  Discontinuation of trastuzumab due to treatment-related TEAE | 1 | 1
  Discontinuation of trastuzumab due to trastuzumab-related TEAE | 0 | 0

8. Secondary Outcome: Number of Participants With AEs Resulting in Dose Modification: Interim Analysis
Description: Dose modification included dose reduction and dose withheld by investigator due to AEs. Dose holds were defined as any instances where planned administration of the study drug was temporarily withheld or interrupted at the direction of the treating physician. Dose reductions of trastuzumab were not allowed; if trastuzumab could not be restarted after being held for a TEAE, it was discontinued.
Time Frame: Up to 49.3 months
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B) | Tucatinib Pre-Crossover (Cohort C)
Number analyzed (Participants) | 86 | 30
Participants
  Tucatinib dose held | 20 | 3
  Tucatinib dose reduced | 8 | 1
  Trastuzumab dose held | 24 | NA — Tucatinib monotherapy arm.
  Trastuzumab infusion interrupted (received full dose within 24 hrs) | 6 | NA — Tucatinib monotherapy arm.
  Trastuzumab infusion stopped early (full dose not received) | 1 | NA — Tucatinib monotherapy arm.

9. Secondary Outcome: Number of Participants With AEs Resulting in Dose Modification: Final Analysis
Description: Dose modification included dose reduction and dose withheld by investigator due to AEs. Dose holds were defined as any instances where planned administration of the study drug was temporarily withheld or interrupted at the direction of the treating physician. Dose reductions of trastuzumab were not allowed; if trastuzumab could not be restarted after being held for a TEAE, it was discontinued. Drug interruption included infusion interrupted (full dose received within 24hrs).
Time Frame: Up to 65.1 months
Population: The safety analysis set included participants who received any amount of study treatment. Data for cohorts A and B was combined as prespecified in SAP.
Measure: Count of Participants; unit: Participants
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B) | Tucatinib Post-Crossover (Cohort C)
Number analyzed (Participants) | 86 | 28
Participants
  Tucatinib dose held | 23 | 7
  Tucatinib dose reduced | 9 | 2
  Trastuzumab dose held | 27 | 2
  Trastuzumab infusion interrupted | 6 | 0

10. Secondary Outcome: Number of Participants With Treatment-Emergent Laboratory Abnormalities (Hematology): Interim Analysis
Description: The following hematology laboratory parameters were assessed: Hemoglobin decreased; leukocytes decreased; neutrophils decreased and Platelets decreased. Treatment emergent laboratory abnormalities were defined as abnormalities that were new or worsened on or after receiving the first dose of study treatment and up through 30 days after the last dose of study treatment. NCI CTCAE v4.03 was used for the lab parameters. Grade 1: mild; Grade 2: moderate; Grade 3: severe or clinically significant; Grade 4: life-threatening.
Time Frame: Up to 49.3 months
Population: The safety analysis set included all participants who received any amount of study treatment. Data for cohorts A and B was combined as prespecified in SAP. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B) | Tucatinib Pre-Crossover (Cohort C)
Number analyzed (Participants) | 85 | 29
Participants
  Hemoglobin decreased, Grade 1 | 28 | 6
  Hemoglobin decreased, Grade 2 | 8 | 2
  Hemoglobin decreased, Grade 3 | 3 | 0
  Hemoglobin decreased, Grade 4 | 0 | 0
  Leukocytes decreased, Grade 1 | 14 | 3
  Leukocytes decreased, Grade 2 | 5 | 0
  Leukocytes decreased, Grade 3 | 0 | 0
  Leukocytes decreased, Grade 4 | 0 | 0
  Neutrophils decreased, Grade 1 | 6 | 1
  Neutrophils decreased, Grade 2 | 2 | 1
  Neutrophils decreased, Grade 3 | 0 | 0
  Neutrophils decreased, Grade 4 | 0 | 0
  Platelets decreased, Grade 1 | 11 | 1
  Platelets decreased, Grade 2 | 2 | 2
  Platelets decreased, Grade 3 | 0 | 0
  Platelets decreased, Grade 4 | 0 | 0

11. Secondary Outcome: Number of Participants With Treatment-Emergent Laboratory Abnormalities (Hematology): Final Analysis
Description: The following hematology laboratory parameters were assessed: Hemoglobin decreased; hemoglobin increased; leukocytes decreased; lymphocytes decreased; neutrophils decreased and Platelets decreased. Treatment emergent laboratory abnormalities were defined as abnormalities that were new or worsened on or after receiving the first dose of study treatment and up through 30 days after the last dose of study treatment. NCI CTCAE v4.03 was used for the lab parameters. Grade 1: mild; Grade 2: moderate; Grade 3: severe or clinically significant; Grade 4: life-threatening.
Time Frame: Up to 65.1 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B) | Tucatinib Post-Crossover (Cohort C)
Number analyzed (Participants) | 85 | 28
Participants
  Hemoglobin decreased, All grades | 42 | 9
  Hemoglobin decreased, Grade 3 | 3 | 0
  Hemoglobin decreased, Grade 4 | 0 | 0
  Hemoglobin increased: All grades | 3 | 0
  Hemoglobin increased: Grade 3 | 0 | 0
  Hemoglobin increased: Grade 4 | 0 | 0
  Leukocytes decreased, All grades | 21 | 5
  Leukocytes decreased, Grade 3 | 0 | 0
  Leukocytes decreased, Grade 4 | 0 | 0
  Lymphocytes decreased, All grades | 25 | 11
  Lymphocytes decreased, Grade 3 | 6 | 1
  Lymphocytes decreased, Grade 4 | 0 | 0
  Neutrophils decreased: All grades | 10 | 0
  Neutrophils decreased: Grade 3 | 0 | 0
  Neutrophils decreased: Grade 4 | 0 | 0
  Platelets decreased, All grades | 15 | 4
  Platelets decreased, Grade 3 | 0 | 0
  Platelets decreased, Grade 4 | 0 | 1

12. Secondary Outcome: Number of Participants With Treatment-Emergent Laboratory Abnormalities (Chemistry): Interim Analysis
Description: The following chemistry laboratory parameters were assessed: Potassium increased; potassium decreased; aspartate aminotransferase increased; creatinine increased; alkaline phosphatase increased; total bilirubin increased. Treatment emergent laboratory abnormalities were defined as abnormalities that were new or worsened on or after receiving the first dose of study treatment and up through 30 days after the last dose of study treatment. NCI CTCAE v5.0 was used for creatinine increased. NCI CTCAE v4.03 was used for the other laboratory parameters. Grade 1: mild; Grade 2: moderate; Grade 3: severe or clinically significant; Grade 4: life-threatening.
Time Frame: Up to 49.3 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B) | Tucatinib Pre-Crossover (Cohort C)
Number analyzed (Participants) | 85 | 29
Participants
  Potassium increased, Grade 1 | 5 | 1
  Potassium increased, Grade 2 | 1 | 0
  Potassium increased, Grade 3 | 0 | 1
  Potassium increased, Grade 4 | 0 | 0
  Potassium decreased, Grade 1 | 13 | 3
  Potassium decreased, Grade 2 | 0 | 0
  Potassium decreased, Grade 3 | 1 | 1
  Potassium decreased, Grade 4 | 0 | 0
  Aspartate Aminotransferase increased, Grade 1 | 20 | 6
  Aspartate Aminotransferase increased, Grade 2 | 3 | 0
  Aspartate Aminotransferase increased, Grade 3 | 2 | 2
  Aspartate Aminotransferase increased, Grade 4 | 3 | 0
  Alanine Aminotransferase increased, Grade 1 | 31 | 4
  Alanine Aminotransferase increased, Grade 2 | 4 | 2
  Alanine Aminotransferase increased, Grade 3 | 2 | 2
  Alanine Aminotransferase increased, Grade 4 | 2 | 0
  Creatinine increased, Grade 1 | 38 | 9
  Creatinine increased, Grade 2 | 11 | 0
  Creatinine increased, Grade 3 | 0 | 0
  Creatinine increased, Grade 4 | 0 | 0
  Alkaline Phosphatase increased, Grade 1 | 16 | 4
  Alkaline Phosphatase increased, Grade 2 | 4 | 2
  Alkaline Phosphatase increased, Grade 3 | 1 | 0
  Alkaline Phosphatase increased, Grade 4 | 0 | 0
  Total Bilirubin increased, Grade 1 | 14 | 6
  Total Bilirubin increased, Grade 2 | 5 | 0
  Total Bilirubin increased, Grade 3 | 3 | 0
  Total Bilirubin increased, Grade 4 | 2 | 0

13. Secondary Outcome: Number of Participants With Treatment-Emergent Laboratory Abnormalities (Chemistry): Final Analysis
Description: The following chemistry laboratory parameters were assessed: Potassium increased; potassium decreased; aspartate aminotransferase increased; creatinine increased; alkaline phosphatase increased; total bilirubin increased; albumin decreased; calcium corrected for albumin decreased; calcium corrected for albumin increased; glomerular filtration rate (GFR), estimated decreased; glucose decreased; glucose increased; sodium decreased; sodium increased; calcium and ionized increased. Treatment emergent laboratory abnormalities: Abnormalities that were new or worsened on or after receiving the first dose of study treatment and up through 30 days after the last dose of study treatment. NCI CTCAE v5.0 used for creatinine increased. NCI CTCAE v4.03 used for the other laboratory parameters. Grade 1: mild; Grade 2: moderate; Grade 3: severe or clinically significant; Grade 4: life-threatening.
Time Frame: Up to 65.1 months
Population: The safety analysis set included all participants who received any amount of study treatment. Data for cohorts A and B was combined as prespecified in SAP. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies number evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B) | Tucatinib Post-Crossover (Cohort C)
Number analyzed (Participants) | 85 | 28
Participants
  Potassium increased, All grades | 6 | 4
  Potassium increased, Grade 3 | 0 | 0
  Potassium increased, Grade 4 | 0 | 0
  Potassium decreased, All grades | 15 | 4
  Potassium decreased, Grade 3 | 1 | 0
  Potassium decreased, Grade 4 | 0 | 0
  Aspartate Aminotransferase increased, All grades | 29 | 9
  Aspartate Aminotransferase increased, Grade 3 | 2 | 3
  Aspartate Aminotransferase increased, Grade 4 | 3 | 0
  Alanine Aminotransferase increased, All grades | 39 | 7
  Alanine Aminotransferase increased, Grade 3 | 2 | 2
  Alanine Aminotransferase increased, Grade 4 | 2 | 0
  Creatinine increased, All grades | 50 | 10
  Creatinine increased, Grade 3 | 0 | 0
  Creatinine increased, Grade 4 | 0 | 0
  Alkaline Phosphatase increased, All grades | 21 | 3
  Alkaline Phosphatase increased, Grade 3 | 1 | 0
  Alkaline Phosphatase increased, Grade 4 | 0 | 0
  Total Bilirubin increased, All grades | 25 | 4
  Total Bilirubin increased, Grade 3 | 3 | 0
  Total Bilirubin increased, Grade 4 | 2 | 0
  Albumin decreased, All grades | 23 | 8
  Albumin decreased, Grade 3 | 1 | 0
  Albumin decreased, Grade 4 | 0 | 0
  Calcium Corrected for Albumin decreased, All grades: number analyzed (Participants) | 84 | 28
  Calcium Corrected for Albumin decreased, All grades | 11 | 5
  Calcium Corrected for Albumin decreased, Grade 3: number analyzed (Participants) | 84 | 28
  Calcium Corrected for Albumin decreased, Grade 3 | 0 | 0
  Calcium Corrected for Albumin decreased, Grade 4: number analyzed (Participants) | 84 | 28
  Calcium Corrected for Albumin decreased, Grade 4 | 0 | 0
  Calcium Corrected for Albumin increased, All grades: number analyzed (Participants) | 84 | 28
  Calcium Corrected for Albumin increased, All grades | 8 | 5
  Calcium Corrected for Albumin increased, Grade 3: number analyzed (Participants) | 84 | 28
  Calcium Corrected for Albumin increased, Grade 3 | 0 | 0
  Calcium Corrected for Albumin increased, Grade 4: number analyzed (Participants) | 84 | 28
  Calcium Corrected for Albumin increased, Grade 4 | 0 | 0
  Glomerular Filtration Rate, Estimated decreased, All grades: number analyzed (Participants) | 77 | 21
  Glomerular Filtration Rate, Estimated decreased, All grades | 51 | 6
  Glomerular Filtration Rate, Estimated decreased, Grade 3: number analyzed (Participants) | 77 | 21
  Glomerular Filtration Rate, Estimated decreased, Grade 3 | 6 | 0
  Glomerular Filtration Rate, Estimated decreased, Grade 4: number analyzed (Participants) | 77 | 21
  Glomerular Filtration Rate, Estimated decreased, Grade 4 | 0 | 0
  Glucose decreased, All grades | 10 | 1
  Glucose decreased, Grade 3 | 0 | 0
  Glucose decreased, Grade 4 | 0 | 0
  Glucose increased, All grades | 48 | 9
  Glucose increased, Grade 3 | 2 | 0
  Glucose increased, Grade 4 | 0 | 0
  Sodium decreased, All grades | 18 | 1
  Sodium decreased, Grade 3 | 5 | 0
  Sodium decreased, Grade 4 | 0 | 0
  Sodium increased, All grades | 7 | 4
  Sodium increased, Grade 3 | 0 | 0
  Sodium increased, Grade 4 | 0 | 0
  Calcium, Ionized increased: All grades: number analyzed (Participants) | 3 | 28
  Calcium, Ionized increased: All grades | 2 | 0
  Calcium, Ionized increased: Grade 3: number analyzed (Participants) | 3 | 28
  Calcium, Ionized increased: Grade 3 | 0 | 0
  Calcium, Ionized increased: Grade 4: number analyzed (Participants) | 3 | 28
  Calcium, Ionized increased: Grade 4 | 0 | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs: Final Analysis
Description: Vital signs included temperature, oxygen saturation, systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate and weight. Vital signs were considered clinically significant: temperature: >= 38 degree Celsius (C); oxygen saturation less than (<)88%; SBP >=120 millimeters of mercury (mmHg) or DBP >=80 mmHg; SBP >=140 mmHg or DBP >=90 mmHg; SBP >=160 mmHg or DBP >=100 mmHg and heart rate >100 beats per minute (bpm) and maximum decrease from baseline in weight in kilograms (kg).
Time Frame: Up to 65.1 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B) | Tucatinib Post-Crossover (Cohort C)
Number analyzed (Participants) | 86 | 28
Participants
  Temperature >=38 degree C | 1 | 0
  Oxygen saturation <88% | 8 | 0
  SBP >= 120 mmHg or DBP >= 80 mmHg | 80 | 27
  SBP >= 140 mmHg or DBP >= 90 mmHg | 49 | 13
  SBP >= 160 mmHg or DBP >= 100 mmHg | 21 | 4
  Heart rate > 100 bpm | 26 | 5
  Maximum decrease from baseline in weight (kg) | 65 | 23

ADVERSE EVENTS:
Time Frame: All-cause mortality: From start of study treatment to death by any cause (maximum up to 71.8 months); adverse events were followed during the safety reporting period (from Day 1 through 30 days after the last dose of study treatment) maximum up to 65.1 months
Description: Adverse events (AEs) for Cohorts A and B were analyzed together as prespecified in SAP. All-Cause Mortality is reported for all enrolled participants, regardless of whether or not they received study drug. SAEs and non-serious AEs are reported only for those participants who received at least one dose of study drug.
Arm/Group | Tucatinib+Trastuzumab (Cohorts A+B) | Tucatinib Pre-Crossover (Cohort C) | Tucatinib Post-Crossover (Cohort C)
All-Cause Mortality (participants affected / at risk) | 54/86 | 2/31 | 15/28
Serious Adverse Events (participants affected / at risk) | 20/86 | 3/30 | 6/28
Other Adverse Events (participants affected / at risk) | 82/86 | 28/30 | 23/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tucatinib+Trastuzumab (Cohorts A+B) (N=86) | Tucatinib Pre-Crossover (Cohort C) (N=30) | Tucatinib Post-Crossover (Cohort C) (N=28)
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Rectal perforation (Gastrointestinal disorders) | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Anorectal infection (Infections and infestations) | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tucatinib+Trastuzumab (Cohorts A+B) (N=86) | Tucatinib Pre-Crossover (Cohort C) (N=30) | Tucatinib Post-Crossover (Cohort C) (N=28)
Anaemia (Blood and lymphatic system disorders) | 9 | 3 | 3
Lacrimation increased (Eye disorders) | 1 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 11 | 6 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2 | 2
Constipation (Gastrointestinal disorders) | 12 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 57 | 10 | 11
Flatulence (Gastrointestinal disorders) | 3 | 1 | 2
Nausea (Gastrointestinal disorders) | 29 | 5 | 2
Oral pain (Gastrointestinal disorders) | 0 | 0 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 2
Vomiting (Gastrointestinal disorders) | 14 | 2 | 4
Asthenia (General disorders) | 3 | 5 | 2
Chills (General disorders) | 16 | 0 | 2
Fatigue (General disorders) | 37 | 6 | 3
Influenza like illness (General disorders) | 7 | 0 | 1
Oedema peripheral (General disorders) | 7 | 2 | 2
Pyrexia (General disorders) | 18 | 3 | 6
COVID-19 (Infections and infestations) | 6 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 4 | 4 | 4
Infusion related reaction (Injury, poisoning and procedural complications) | 18 | 0 | 4
Alanine aminotransferase increased (Investigations) | 5 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 5 | 3 | 3
Ejection fraction decreased (Investigations) | 5 | 0 | 1
Weight decreased (Investigations) | 8 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 17 | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 7 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 1 | 6
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 2 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 1 | 1
Dizziness (Nervous system disorders) | 5 | 2 | 1
Dysgeusia (Nervous system disorders) | 4 | 1 | 1
Headache (Nervous system disorders) | 9 | 3 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 1 | 0
Anxiety (Psychiatric disorders) | 9 | 0 | 0
Insomnia (Psychiatric disorders) | 7 | 1 | 0
Dysuria (Renal and urinary disorders) | 3 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 17 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 2 | 1
Hypertension (Vascular disorders) | 15 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 1
Blepharospasm (Eye disorders) | 2 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 3 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 4 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 2 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1
Noninfective gingivitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 3 | 0 | 0
Pain (General disorders) | 2 | 0 | 0
Peripheral swelling (General disorders) | 2 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gingival abscess (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 0 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 1
Influenza (Infections and infestations) | 2 | 0 | 0
Nail infection (Infections and infestations) | 3 | 0 | 1
Otitis media (Infections and infestations) | 2 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 0 | 0
Blood creatinine increased (Investigations) | 4 | 0 | 1
Weight increased (Investigations) | 3 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neurotoxicity (Nervous system disorders) | 0 | 1 | 1
Restless legs syndrome (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 1
Haematuria (Renal and urinary disorders) | 4 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 4 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 4 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 2 | 0
Eructation (Gastrointestinal disorders) | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Pregnancy of partner (Social circumstances) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/13/NCT03043313/Prot_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT03043313/SAP_001.pdf
  • Statistical Analysis Plan: Addendum (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT03043313/SAP_003.pdf